CLINICAL TRIAL: NCT02298686
Title: Biomarker for Sanfilippo Disease Type A-B-C-D AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Biomarker for Sanfilippo Type A-B-C-D Disease (BioSanfilippo)
Acronym: BioSanfilippo
Status: Withdrawn | Type: Observational
Why Stopped: Transition to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BSF01-2014
Record Dates: First submitted 2014-10-23; First posted 2014-11-24 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Mental Retardation; Developmental Delay
Keywords: Sanfilippo Disease Type A-B-C-D; Biomarker
MeSH Terms: conditions — Intellectual Disability; Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectrometry 10 ml EDTA blood or a dry blood spot filter card are taken. To proof the correct Sanfilippo Type A-B-C-D diagnosis in those patients where up to the enrollment in the study no ge-netic testing has been done, sequencing of Sanfilippo Type A-B-C-D will be done. The analyses will be done at the:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Sanfilippo Type A-B-C-D disease or high-grade suspicion for Sanfilippo Type A-B-C-D disease

SUMMARY:
Development of a new MS-based biomarker for the ear-ly and sensitive diagnosis of Sanfilippo Disease Type A-B-C-D from blood (plasma)

DETAILED DESCRIPTION:
The Mucopolysaccharidoses (MPS Disorders) are a group of rare genetic disorders caused by the deficiency of one of the lysosomal enzymes, resulting in an inability to metabolize complex carbohydrates (mucopolysaccharides) into simpler molecules. High concentrations of mucopolysaccharides in the cells of the central nervous system, including the brain, cause the neu-rological and developmental deficits that accompany these disorders.

Lysosomal enzymes are found in the lysosome, a very small membrane-contained body (organelle) found in the cytoplasm of most cells. The lysosome is often called the "waste disposal plant" of the cell. The accumulation of these large, undegraded mucopolysaccharides in the cells of the body is the cause of a number of physical symptoms and abnormalities.

MPS-III (Sanfilippo Syndrome) is one of seven MPS Disorders. It is an inborn error of metabolism that is transmitted as an autosomal recessive genetic disorder. MPS-lll has been categorized into four subtypes: MPS-III Type A, MPS-III Type B, MPS-III Type C, and MPS-III Type D depending on the gene defect (MPS3A - SGSH gene, MPS3B - NAGLU gene, MPS3C - HGSNAT, MPS3D - GNS gene). All types are associated with some degree of mental deterioration, but the severity depends on the particular type of MPS-lll. Several physical defects may be present, and the severity of these defects varies with the type of MPS-III. In the case of each type of MPS-III, abnormal amounts of a specific, chemically complex molecule is excreted in the urine. The excreted chemical is the same for each of the four types of MPS-III, since the defective gene involves a different step, and thus a different enzyme, in the deconstruction of the same mucopolysaccharide. By testing for one or another of these enzymes, the variant type may be readily identified.

Symptoms Patients with Sanfilippo Syndrome (MPS Type III) usually appear normal at birth, but mental retardation and developmental delay is usually evident by age 3-5 years. Mental and motor development reaches a peak by 3-6 years of age after which behavioral disturbances and intellectual decline usually occur. However, hyperactivity and irritability may become obvious earlier.

The following symptoms are usually apparent by approximately age 10: neurological deficits and signs, wobbly and erratic gait and difficulty walking (ataxia), hyperactivity (hyperkinetic syndrome), mental retardation, stiff joints, hernias, enlarged liver and/or spleen (hepatosplenomegaly).Growth is usually minimally affected; the head may be enlarged, and abnormal hairiness (hirsutism) may occur. Mild coarsening of facial features also characterizes this disorder. In some cases deafness may also occur.

Causes All four varieties of MPS-III are autosomal recessive genetic disorders.

The gene abnormalities associated with MSS-IIIA, MPS-IIIB, MPS-IIIC and MPS-IIID have been identified. The Gene Map Loci are as follows:

MPS-IIIA --------- 17q25.3; SGSH gene

MPS-IIIB --------- 17q21.2; NAGLU gene

MPS-IIIC --------- 8p11.21; HGSNAT gene

MPS-IIID --------- 12q14.3; GNS gene

Genetic diseases are determined by the combination of genes for a particular trait that are on the chromosomes received from the father and the mother.

Recessive genetic disorders occur when an individual inherits the same abnormal gene for the same trait from each parent. If an individual receives one normal gene and one gene for the disease, the person will be a carrier for the disease, but usually will not show symptoms. The risk for two carrier parents to both pass the defective gene and, therefore, have an affected child is 25% with each pregnancy. The risk to have a child who is a carrier like the parents is 50% with each pregnancy. The chance for a child to receive normal genes from both parents and be genetically normal for that particular trait is 25%. The risk is the same for males and females.

All individuals carry 4-5 abnormal genes. Parents who are close relatives (consanguineous) have a higher chance than unrelated parents to both carry the same abnormal gene, which increases the risk to have children with a recessive genetic disorder.

ELIGIBILITY:
INCLUSION CRITERIA:

* Informed consent will be obtained from the patient or the parents before any study related procedures.
* Patients of both genders older than 2 month
* The patient has a diagnosis of Sanfilippo Type A-B-C-D disease or a high-grade suspicion for Sanfilippo Type A-B-C-D disease
* High-grade suspicion present, if one or more inclusion criteria are valid:

  * Positive family anamnesis for Sanfilippo Type A-B-C-D disease
  * Dysostosis multiplex without identifiable cause
  * Splenomegaly without identifiable cause
  * Hepatomegaly without identifiable cause
  * Heparan sulfate excretion in urine
  * CNS involvement without identifiable cause

EXCLUSION CRITERIA:

* No Informed consent from the patient or the parents before any study related procedures.
* Patients of both gender younger than 2 month
* No diagnosis of Sanfilippo Type A-B-C-D disease or no valid criteria for profound suspicion of Sanfilippo Type A-B-C-D disease

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Sanfilippo Type A-B-C-D disease or high-grade suspicion for Sanfilippo Type A-B-C-D disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Sanfilippo Type A-B-C-D disease from plasma | 24 months
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker | 36 months
  the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (5):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided